CLINICAL TRIAL: NCT06618222
Title: An Ambispective, Multicenter Clinical Study to Evaluate the Safety and Efficacy of the Wingspan Stent System for Clinical Use
Brief Title: Wingspan Stent System for Intracranial Artery Stenosis
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Other Study IDs: Wingspan PMS
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Artery Stenosis; Stent; Endovascular Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wingspan stent: All patients had received Percutaneous transluminal angioplasty and stenting with Wingspan stent system.
  Interventions: Device: Wingspan stent system

INTERVENTIONS:
Device: Wingspan stent system — All patients had received Percutaneous transluminal angioplasty and stenting with Wingspan stent system.

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of Wingspan Stent System in "real world" patients with intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
This study is an ambispective, multicenter clinical study design and consecutively included patients with symptomatic intracranial atherosclerotic arterial stenosis (stenosis rate of 70%-99%) with the Wingspan stent system between December 2022 and June 2023.

All included patients underwent preoperative DSA to clarify the diagnosis, and were followed up within 6 months after the procedure with DSA to clarify in-stent restenosis. The main observations endpoints included revascularization within 30 days after the procedure, revascularization within 31 days to 6 months, symptomatic in-stent restenosis within 6 months after the procedure, stroke or death within 30 days or ischaemic stroke in the qualifying artery beyond 30 days through 6 months, stroke (ischaemic or hemorrhagic stroke) or death in the qualifying artery within 30 days, ischaemic stroke that occurs beyond the lesion arterial territory from 31 days to 6 months after the procedure, any cerebral parenchymal hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage from 31 days to 6 months after the procedure, all-cause death (cerebrovascular death and non-cerebrovascular death) from 31 days to 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 80 years of age;
2. Patients with symptomatic intracranial atherosclerotic stenosis who failed antiplatelet therapy or poor collateral circulation compensation or hypoperfusion in the territory of the culprit artery;
3. Digital Subtraction Angiography(DSA) showed 70% to 99% stenosis in target intracranial artery;
4. The target lesion was in the internal carotid artery (intracranial segment), middle cerebral artery, vertebral artery (intracranial segment), basilar artery, and it was a single lesion that required surgical treatment;
5. The patient voluntarily underwent treatment with the Wingspan stent system;
6. mRS < 3 (if any);
7. The onset of the latest transient ischemic attack (TIA) was not limited or ischemic stroke occurred within 2 weeks prior to stenting procedure;
8. Willingness to participate in this clinical trial and signing the consent form, and be able to complete the corresponding inspections, follow ups, etc. according to the requirements of the clinical protocol during the clinical trial.

Exclusion Criteria:

1. The target vessels was complete occlusion;
2. >70% stenosis observed at the intracranial large-vessel distal to the target vessel or >70% stenosis observed at the intracranial/extracranial large-vessel proximal to the target vessel;
3. Preoperative magnetic resonance showed perforating infarction in the target lesion area;
4. Preoperative CT showed that there was hemorrhage transformation after infarction in the target vessel area, or a history of primary cerebral hemorrhage, or a history of subarachnoid, subdural and epidural hemorrhage within 30 days before operation, or there was no treatment Chronic subdural hematoma ≥5mm;
5. Hospitalized surgical treatment within 30 days before operation, or planned hospitalized surgical treatment within 6 months after surgery;
6. CT showed Severe calcified lesions;
7. Previously received endovascular treatment or surgical intervention at the target vessel (except for patients with simple balloon dilatation);
8. Non-atherosclerosis lesions;
9. Patients with potential sources of cardiac embolism (such as atrial fibrillation, left ventricular thrombosis, myocardial infarction within 6 weeks);
10. Concomitant intracranial tumor, aneurysm or intracranial arteriovenous malformation;
11. Known hypersensitivity to aspirin, heparin, clopidogrel, rapamycin (sirolimus), lactic acid polymer, poly-n-butyl methacrylate, nickel-titanium alloy, or contraindications to anesthetics and contrast agents;
12. Hemoglobin <100g/L, platelet count <100*109/L, International normalized ratio (INR) >1.5 (irreversible) or uncorrectable hemorrhagic factors;
13. Uncontrollable severe hypertension (systolic blood pressure>180 millimetres of mercury (mmHg) or diastolic blood pressure>110mmHg);
14. Known liver or renal insufficiency (aspartate transaminase (ALT)> 3x upper limit or aspartate transaminase > 3x upper limit, Serum creatinine#250μmol/L);
15. Life expectancy < 1 year;
16. Pregnant/lactating female patients;
17. Patients with cognitive impairment or mental diseases (except for those with cognitive impairment due to arterial stenosis);
18. Patients who were participated in other clinical trials within 3 months or participating in other clinical trials who had not yet reached the primary clinical endpoint.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: symptomatic ICAS (stenosis rate of 70%-99%) with the Wingspan stent system between December 2022 and June 2023
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
The incidence of In-stent restenosis within 6 months after operation | 6 months after operation
  In-Stent Restenosis (ISR) is defined as stenosis greater than 50% within or immediately adjacent (within 5 mm) to the implanted stents and absolute luminal loss greater than 20% at 6 months follow-up imaging.

SECONDARY OUTCOMES:
Stent success / Procedure success | Immediately after operative
  Stent success is defined as Wingspan is successfully implanted into the vascular site of the target lesion with balloon pretreatment and the delivery system was successfully withdrawn.
  Procedure success is defined as a reduction in the degree of stenosis to ≤ 30% after the application of any interventional treatment method.
Rate of good functional outcomes measured by Modified Rankin Score (mRS) | 30days, 6 months after operation
  Modified rankin score measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The range is 0-6 (0 is highest function with no symptoms and 6 is death). This outcome measured percentage of subjects with a "good"; functional outcome with a score ranging from 0-2.
Percent of Participants With National Institutes of Health Stroke Scale (NIHSS) Score = 0 or 1 at 6 months follow-up | 6 months after operation
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).
Rate of all revascularization and target lesion revascularization | 30days, 31days to 6 months after operation
  The proportion of patients who had revascularization in target lesion or not.
Symptomatic ISR within 6 months | within 6 months
  Symptomatic ISR is defined as ISR associated with ischemic event in the territory.
Any stroke or death within 30 days after operation, and the incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months after operation. | 30days, 31days to 6 months after operation
  As a composite endpoint include any stroke or death within 30 days, and the incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months after operation.
Any stroke or death within 30 days after operation | Within 30days after operation
  Any stroke, death means death from any cause, including stroke or cerebrovascular disease.
Stroke (including hemorrhage or ischemic stroke) or death within 30 days associated with the target vessel | Within 30days after operation
  The proportion of patients who had any stroke or died within 30 days after operation in association with stenting implantation.
The incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months after operation | 31days to 6 months after operation
  There is clear imaging evidence to confirm that the target vessel area is occluded again, which leads to ischemic stroke.
The incidence of recurrent ischemic stroke outside the target vascular area within 31 days to 6 months after operation | 31days to 6 months after operation
  There is clear imaging evidence to confirm that outside the target vessel area is occluded again, which leads to ischemic stroke.
Any parenchymal hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage | 31days to 6 months after operation
  There is clear imaging evidence to confirm that the incidence of any parenchymal hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage.
All cause death | 31days to 6 months after operation
  The proportion of patients who died from all causes is evaluated from 31 days to 6 months after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Ya Deng, Principal Investigator — The First People's Hospital of Changzhou
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China